CLINICAL TRIAL: NCT06277609
Title: Interventional, Open-label, Repeated Single-dose Trial Investigating the Effects of Enzyme Inhibition on the Pharmacokinetic Profile of Lu AF28996 and Its Metabolites in Healthy Participants
Brief Title: A Trial Investigating Lu AF28996 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20508A
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Aspirin; Mefenamic Acid; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Lu AF28996 with Enzyme Inhibitors (Experimental): Participants will receive repeated single doses of Lu AF28996 and enzyme inhibitors.
  Interventions: Drug: Lu AF28996; Drug: Acetylsalicylic Acid; Drug: Mefenamic Acid
- Part B: Lu AF28996 with Antibiotics (Experimental): Participants will receive single doses of Lu AF28996 and amoxicillin/clavulanic acid.
  Interventions: Drug: Lu AF28996; Drug: Amoxicillin/clavulanic acid

INTERVENTIONS:
Drug: Lu AF28996 — Capsule
Drug: Acetylsalicylic Acid — Tablet
  Arms: Part A: Lu AF28996 with Enzyme Inhibitors
Drug: Mefenamic Acid — Tablet
  Arms: Part A: Lu AF28996 with Enzyme Inhibitors
Drug: Amoxicillin/clavulanic acid — Tablet
  Arms: Part B: Lu AF28996 with Antibiotics

SUMMARY:
The purpose of this study is to investigate repeated doses of Lu AF28996 in healthy participants and co-administered with two other compounds, and in a separate cohort following co-administration with antibiotics, to see how well the doses are tolerated and what the body does to the drug after administering it.

DETAILED DESCRIPTION:
The study has 2 parts: Part A and Part B.

Part A will consist of 2 cohorts (Cohorts A1 to A2), with 8 participants per cohort and will receive single doses of Lu AF28996 alone and in combination with enzyme inhibitors.

Part B will consist of one cohort (Cohort B1), with 8 participants who will all receive single doses of Lu AF28996 alone and in combination with amoxicillin/clavulanic acid.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤30 kilograms per meter squared (kg/m^2) at the Screening Visit and at the Safety Baseline Visit.
* The participant has a resting supine pulse ≥50 and ≤100 beats per minute (bpm) at the Screening Visit and at the Safety Baseline Visit.
* The participant has a resting supine systolic blood pressure ≥90 and ≤140 millimeters of mercury (mmHg) and a resting supine diastolic blood pressure ≥50 and ≤90 mmHg at the Screening Visit and at the Safety Baseline Visit.
* The participant has a normal circadian rhythm, defined as a person who usually wakes between 6:00 and 9:00 a.m. and goes to sleep between 9:00 p.m. and midnight.

Exclusion Criteria:

* The participant is a member of the site staff or of their immediate families or is a subordinate (or immediate family member of a subordinate) to any of the site staff.
* Part B only, the participant is a woman of childbearing potential AND is using oral hormonal contraceptives.
* The participant has previously been enrolled in this trial.
* The participant has previously been dosed with Lu AF28996.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-05-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Lu AF28996 | Predose to Day 13
Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Lu AF28996 | Predose to Day 13

SECONDARY OUTCOMES:
Nominal Time Corresponding to the Occurrence of Cmax | Predose to Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Dallas CRU, Dallas, Texas, United States